CLINICAL TRIAL: NCT04768049
Title: Cross-cultural Translation and Validity of the Pediatric Balance Scale (PBS) Into Urdu.
Brief Title: Urdu Version of Pediatric Balance Scale
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/00746 Saima Mahmood
Record Dates: First submitted 2021-02-18; First posted 2021-02-24 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Cerebral Palsy
Keywords: Pediatric Balance scale; Cerebral palsy; Urdu version
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tool Translation — Data Collection procedure will be done in two phases. The first phase will revolve around the translation of the instrument. Firstly the tool will be translated into Urdu with help of two professional translators and then it will be back translated into English to cross check the clarity of text. The translation will focus more on the context and understanding of the text rather literal word-to-word meanings. The translation will be done according to the WHO guidelines

SUMMARY:
Children with cerebral palsy often suffer from a lack of balance compared with typically developing children. Because balance capacity is relevant to functional activities, reliable and valid functional balance measures are crucial for the pediatric clinical setting in local native languages, so the aim of this study is to translate the Pediatric Balance Scale (PBS) into Urdu and to find the reliability and validity of the translated version Pediatric Balance Scale (PBS) in cerebral palsy.

DETAILED DESCRIPTION:
Cross cultural researches are scientific methods which focus on making systematic comparisons from culture to culture responding to questions about the reasons of occurrence, dissemination and sources of variety in different cultures about compound issues referring to a similar problem across the globe arising from a wide spread field e.g. language which is an integral part of culture . Children with cerebral palsy often suffer from a lack of balance compared with typically developing children. Because balance capacity is relevant to functional activities, reliable and valid functional balance measures are crucial for the pediatric clinical setting.

Cerebral palsy is the most commonly affecting physical dysfunction of childhood. In United States alone 9200 - 9500 children including both infants and preschools are labelled with Cerebral palsy on yearly basis. It has a variety of appearances from isolated to global mental and mental impairments causing disturbance in a multiplicity of motor and cognitive functions such as gait disturbance and cognitive issues.

There are a lot of tools available which are used in physical therapy to assess balance in adults as well as children living with cerebral palsy and out of these tools one commonly used tool for pediatric population is Pediatric Balance Scale (PBS). According to the ICF domain it lies in the "Activity" category. The primary purpose of this scale is to evaluate and discriminate the capacity to maintain and achieve balance both in sitting and standing positions. It is a 14- item questionnaire, takes less than 15 minutes to administer and is used for cerebral palsy population aged between 5-15 years. In clinical settings standardized tools are thought useful in attaining scholarly objectives. But these standardized tools don't seem to serve their purpose to the fullest specifically in situations when they become indifferent to the culture and language of the population they are addressed to. This ultimately makes the assessment of persons from a varied culture groups difficult and hence makes the need of translations significant.

According to the reviewed literature Pediatric Balance Scale has already been translated into many other languages like Brazilian, Persian and Turkish. Validity and reliability of the tool has also been established in the fore mentioned languages. Despite being the need, till date Pediatric Balance Scale has not been translated into Urdu language. This study targets at the cross cultural adaptation of the tool's contents and the evaluation of the face validity, content validity, discriminate validity, construct validity, internal consistency and reliability of the translated version of pediatric balance scale will also be done for children diagnosed with Cerebral Palsy falling in the inclusion criteria.

In 2012 Lilian G K Ries conducted a research along with the research mates at University of Estado de Santa Catarina, Brazil under the title of "Cultural-adaptation and Reliability analysis of Brazilian version of pediatric balance scale (PBS)" and the results of this study concluded that PBS is adequately reliable for children diagnosed with Cerebral Palsy and having GMFCS level I and II. In 2019, Elnaz ALIMIl et al conducted a study with the aim to evaluate the Test-retest and inter-rater reliability of Persian version of Pediatric Balance Scale in children with spastic Cerebral Palsy. They concluded the study with the notion that the PBS shows high inter-rater reliability & the test-retest reliability appropriate for measuring functional balance in children with spastic cerebral palsy with mild to moderate motor impairment. Arzu Erden conducted a study in 2020 to evaluate the Reliability and validity of Turkish version of PBS and showed that the Turkish version of the scale is a valid and reliable tool to evaluate children with balance impairments.

Another study conducted by Gi-won kim et al in 2010 evaluated reliability of PBS based on raters clinical experience and test experience showed high inter rater and intra rater reliability. In 2012 Jin Gang Her's study on Reliability of Pediatric Balance Scale in assessment of the children with cerebral palsy showed high inter rater and intra rater reliability of Pediatric Balance Scale in Children with Cerebral Palsy.In 2017 Sivatejaa Panibatla's study on Relationship of trunk control and balance in children with cerebral palsy suggested a strong correlation between trunk control and balance when evaluated using PBS.

In 2013 Mary rose et al showed in her study about the pediatric balance scale: a modified version of the berg scale for children with mild to moderate motor impairment that PBS demonstrate good test-retest and interrater reliability when used with school-age children with mild to moderate motor impairments.In 2000 Palisano et al conducted a study on validation of a model of GMFC in children with CP suggests that distinction between GMFC levels are meaningful. In 2013 Beatriz O et al suggested about Portuguese version of pediatric berg balance scale that this is a reliable tool to be used in balance assessment of Portuguese Children. A study conducted by Sue-mae gan et al in 2008 on psychometric properties of functional balance assessment in children with cerebral palsy and concluded that the 3 functional balance measures are simple, valid, and reliable for examining children with cerebral palsy and are thus suitable for clinical practice

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of spastic hemi and diplegic CP
* age between 5 and 15 years,
* able to accept and follow verbal instructions,
* ability to independently maintain a standing position for at least four seconds,
* Gross Motor Function Classification System [GMFCS] levels I-II)

Exclusion Criteria:

* • Suffering from any other condition that interfered with physical activity.

  * Quadriplegic Flaccid CP, Choreo atheotoid CP

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: • To translate the Pediatric Balance Scale (PBS) into Urdu, and to find the reliability and validity of the translated version Pediatric Balance Scale (PBS) in cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Pediatric balance scale | up to 24 weeks
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MSNMPT, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Pakistan General Railway Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saether R, Helbostad JL, Riphagen II, Vik T. Clinical tools to assess balance in children and adults with cerebral palsy: a systematic review. Dev Med Child Neurol. 2013 Nov;55(11):988-99. doi: 10.1111/dmcn.12162. Epub 2013 May 16. PMID 23679987
- [Background] Mason TC. Cross-cultural instrument translation: assessment, translation, and statistical applications. Am Ann Deaf. 2005 Spring;150(1):67-72. doi: 10.1353/aad.2005.0020. PMID 15969225
- [Background] Ries LG, Michaelsen SM, Soares PS, Monteiro VC, Allegretti KM. Cross-cultural adaptation and reliability analysis of the Brazilian version of Pediatric Balance Scale (PBS). Rev Bras Fisioter. 2012 Jun;16(3):205-15. doi: 10.1590/s1413-35552012005000026. Epub 2012 Jun 14. English, Portuguese. PMID 22699691
- [Background] Erden A, Acar Arslan E, Dundar B, Topbas M, Cavlak U. Reliability and validity of Turkish version of pediatric balance scale. Acta Neurol Belg. 2021 Jun;121(3):669-675. doi: 10.1007/s13760-020-01302-9. Epub 2020 Feb 19. PMID 32077065
- [Background] ALIMIl E, Kalantari M, Nazeri AR, Akbarzade Baghban A. Test-retest & Inter-rater Reliability of Persian Version of Pediatric Balance Scale in Children with Spastic Cerebral Palsy. Iran J Child Neurol. 2019 Fall;13(4):163-171. PMID 31645876
- [Background] Kim G-w. The Reliability of Pediatric Balance Scale on Rater's Clinical work expereience and Test experience The Journal Korean Society of Physical Therapy. 2010.Her J-G. Reliability of Pediatric Balance Scale in Assesment of the Children with Cerebral Palsy 2012;24(301-305).